CLINICAL TRIAL: NCT01025518
Title: A Randomized Trial Evaluating Resistance Training and Dietary Supplements as Intervention for Regaining Muscle Mass Following Radiotherapy in Head and Neck Cancer Patients
Brief Title: DAHANCA 25A: Resistance Training and Dietary Supplements as Intervention for Regaining Muscle Mass Following Radiotherapy in Head and Neck Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Head and Neck Cancer Group (Network)
Collaborators: Danish Center for Interventional Research in Radiation Oncology (CIRRO) (Other)
Responsible Party: Principal Investigator, Jens Overgaard, Professor, MD, Danish Head and Neck Cancer Group
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DAHANCA 25A; CIRRO-IP010309 (Other Grant/Funding Number: CIRRO); Ethical Comittee: 20090181
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Head and Neck Neoplasms
Keywords: Head and Neck Neoplasms; Resistance training; Muscle mass; Functional capacity
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Resistance Training; Proteins; Creatine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- resistance training and dietary supplement (Experimental)
  Interventions: Other: Resistance training; Dietary Supplement: Protein and creatine
- Resistance training and placebo ingestion (Placebo Comparator): 12 weeks of resistance training and placebo ingestion
  Interventions: Other: Resistance training; Dietary Supplement: Placebo

INTERVENTIONS:
Other: Resistance training — 12 weeks of resistance training in combination with protein and creatine or placebo ingestion
Dietary Supplement: Protein and creatine — 30 g of protein with each training session, 5 g of creatine pr day
  Other Names: In2Zyme WP80 and In2Zyme Biodrive 1
  Arms: resistance training and dietary supplement
Dietary Supplement: Placebo — Maltodextrine
  Arms: Resistance training and placebo ingestion

SUMMARY:
The purpose of this study is to investigate whether resistance training in combination with dietary supplementation is tolerable among head and neck cancer patients and to evaluate the possible effect on muscle mass, strength and functional capacity.

DETAILED DESCRIPTION:
Head and neck cancer patients experience a significant loss of muscle mass following radiotherapy treatment due to cachexia and dysphagia. This negatively affects muscle strength and functional capacity.

Studies on healthy individuals and various groups of patients show that resistance training in combination with protein and creatine ingestion is an effective means of increasing muscle mass, strength and functional capacity.

Thus the aim is to investigate the following:

* is resistance training and dietary supplements tolerable among head and neck cancer patients
* the effect of the intervention on muscle mass, strength and functional capacity

ELIGIBILITY:
Inclusion Criteria:

* head and neck cancer patients (localized to the larynx, pharynx and oral cavity) treated with curative radiotherapy
* complete loss of tumor
* WHO performance status between 0-1 and expected ability to complete the training protocol
* No parenteral feeding
* above the age of 18
* written concent

Exclusion Criteria:

* other malignant diseases
* pregnancy
* undergoing systematic resistance training or creatin ingestion
* Alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Muscle mass and muscle strength | 13 weeks

SECONDARY OUTCOMES:
Functional capacity | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jens Overgaard, Professor, MD, Study Chair — DAHANCA
Locations (2):
- Denmark (2):
  - Dept. of Experimental Clinical Oncology, Aarhus University Hospital, Aarhus, Region Midt
  - Dept. of Experimental Clinical Oncology, Aarhus

REFERENCES:
- See also: Danish Head and Neck Cancer Group — http://www.dahanca.dk